CLINICAL TRIAL: NCT06142721
Title: Comparison of Walking Parameters Between Idiopathic Toe Walking Children and Children With Independent Walking Diparetic Cerebral Palsy
Brief Title: Comparison of Walking Parameters Between Idiopathic Toe Walking and Independent Walking Diparetic Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Fatih EROL, Principal Investigator, Biruni University
Other Study IDs: FEROL
Record Dates: First submitted 2023-03-05; First posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Gait Disorders in Children; Cerebral Palsy Spastic Diplegia
Keywords: Toe walking; cerebral palsy; idiopathic toe walking; 3D gait analysis
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ITW Group: 3D gait analysis was applied to children with idiopathic toe walking. Static, kinematic and kinetic walking parameters were evaluated.
  Interventions: Other: 3D Gait Analysis
- DCP Group: 3D gait analysis was applied to diparetic children who were able to walk independently. Static, kinematic and kinetic walking parameters were evaluated.
  Interventions: Other: 3D Gait Analysis
- Healthy Group: 3D gait analysis was applied to healthy children. Static, kinematic and kinetic walking parameters were evaluated.
  Interventions: Other: 3D Gait Analysis

INTERVENTIONS:
Other: 3D Gait Analysis — 3D gait analysis was applied to children. Static, kinematic and kinetic walking parameters were evaluated

SUMMARY:
The aim of the observational study is to compare static, kinematic and kinetic parameters with normal gait parameters in cases with Idiopathic toe walking (ITW) and Diparetic Cerebral Palsy (DCP) who have Gross Motor Function Classification System 1 level with the 3D Gait Analysis method, and to enable the early diagnosis of DCP and ITW. Male and female cases aged between 3-18 years will be included. This study will be carried out at Acıbadem Altunizade Hospital.

DETAILED DESCRIPTION:
It is an observational study. The aim of the observational study is to compare static, kinematic and kinetic parameters with normal gait parameters in cases with Idiopathic toe walking (ITW) and Diparetic Cerebral Palsy (DCP) who have Gross Motor Function Classification System 1 level with the 3D Gait Analysis method, and to enable the early diagnosis of DCP and ITW. Male and female cases aged between 3-18 years will be included. This study will be carried out at Acıbadem Altunizade Hospital. 51 cases will be included in our study. These cases will be divided into three groups. The first group will consist of patients diagnosed with idioaptic toe walking (n:17), the second group will be composed of diparetic cerebral palsy (n:15) with independent ambulation, and the third group will be the control group (n:19). First, the demographic information of the cases will be recorded. With 3D walking analysis, kinetic, kinematic and static data will be collected. The analysis of the obtained data will be done with Polygon Software (Vicon, Oxford, UK). Evaluated kinetic, kinematic and static parameters will be compared between three groups.

Is the lower extremity compensation of children with diparetic cerebral palsy who can walk independently more than children with idiopathic toe walking?

ELIGIBILITY:
Inclusion Criteria:

* Voluntary consent from family
* Diagnosed with idiopathic toe walking and spastic diparesis between the ages of 3-18.
* Cases with GMFCS 1
* The patients who applied to the healthy children's clinic, showed typical development, did not have any musculoskeletal and neurological problems, and wished to voluntarily participate in the study were included in the control group.

Exclusion Criteria:

* Refusing to participate in the study
* Under the age of 3 and over the age of 18
* Not at GMFCS 1 level
* Cases who did not have any orthopedic problems other than accompanying toe walking were excluded from the study.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: A total of 51 cases, including 17 ITW(female:4;male:13), 15 DCP(female:5;male:10) and 19 Control groups (female:6;male:13), were included.
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
3D Gait Analysis | Baseline
  Sixteen markers defined according to the Modified Helen Heyes protocol are applied to certain anatomical regions of both lower extremities. 3D gait analysis can precisely calculate joint angles and movement patterns in all three planes. Collect spatio-temporal data.

CONTACTS AND LOCATIONS:
Overall Officials: Fatih Erol, Principal Investigator — Biruni University
Locations (1):
- Acıbadem Altunizade Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available to other researchers.